CLINICAL TRIAL: NCT02154529
Title: A Phase 1b/2a Study of the Combination of KD019 and Trastuzumab in Subjects With HER2-Positive Metastatic Breast Cancer
Brief Title: Study of the Combination of KD019 and Trastuzumab in Subjects With HER2-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor closed the study due to lack of response.
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD019-204
Record Dates: First submitted 2014-05-28; First posted 2014-06-03 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: HER-2 Positive Breast Cancer; Metastatic Malignant Neoplasm to Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — XL647; Trastuzumab

STUDY DESIGN:
Intervention Model Description: A phase 1b ascending dose-finding study for establishing the maximum tolerated dose (MTD) of tesevatinib (with trastuzumab).
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV (Experimental): Tesevatinib in combination with Trastuzumab: tesevatinib 150 mg PO QD in combination with trastuzumab 8 mg/kg IV initially then 6 mg/kg IV every 3 weeks thereafter.
  Interventions: Drug: Tesevatinib; Drug: Trastuzumab
- Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV (Experimental): Tesevatinib in combination with Trastuzumab: tesevatinib 250 mg PO QD in combination with trastuzumab 8 mg/kg IV initially then 6 mg/kg IV every 3 weeks thereafter.
  Interventions: Drug: Tesevatinib; Drug: Trastuzumab
- Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV (Experimental): Tesevatinib in combination with Trastuzumab: tesevatinib 300 mg PO QD in combination with trastuzumab 8 mg/kg IV initially then 6 mg/kg IV every 3 weeks thereafter.
  Interventions: Drug: Tesevatinib; Drug: Trastuzumab
- Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV (Experimental): Tesevatinib in combination with Trastuzumab: tesevatinib 350 mg PO QD in combination with trastuzumab 8 mg/kg IV initially then 6 mg/kg IV every 3 weeks thereafter.
  Interventions: Drug: Tesevatinib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Tesevatinib
  Other Names: KD019; XL647
Drug: Trastuzumab

SUMMARY:
Evaluate the safety and tolerability and determine the maximum tolerated dose (MTD) of the combination of tesevatinib and trastuzumab in subjects with HER2-positive metastatic breast cancer

DETAILED DESCRIPTION:
This is a multicenter, Phase 1b/2a, multiple ascending-dose, open-label study designed to assess the safety, tolerability, and efficacy of tesevatinib (KD019) in combination with trastuzumab in subjects with human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer. The study planned to include a Phase 2a expansion in which approximately 50 subjects would receive tesevatinib at the maximum tolerated dose (MTD) dose determined in Phase 1b.

The study employs a successive cohort dose-escalation designed to determine the MTD of tesevatinib in combination with trastuzumab. The MTD dose is defined as the dose level below in which : (a) 2 of 3 subjects (or 2 of 6 subjects if Grade ≥ 3 tesevatinib related treatment emergent adverse event [TEAE] experience in 1 of the first 3 subjects).

In the Phase 1b portion of the study, tesevatinib is to be administered orally (PO) to successive cohorts of subjects at 150 mg, 250 mg, 300 mg, 350 mg, and 400 mg once daily (QD).

The following 4 dossing cohorts are initiated during the study:

* Cohort 1: 150 mg tesevatinib PO QD
* Cohort 2: 250 mg tesevatinib PO QD
* Cohort 3: 300 mg tesevatinib PO QD
* Cohort 4: 350 mg tesevatinib PO QD

[Note: the sponsor suspended the study before a cohort of subjects were enrolled at tesevatinib 400 mg PO QD.]

Trastuzumab is administered intravenously (IV) at 8 mg/kg as an initial loading dose on Day 1 of Cycle 1, followed by 6 mg/kg IV every 3 weeks thereafter, beginning Day 1 of Cycle 2. Subjects entering the study already on trastuzumab are not to receive the initial loading dose and instead receive trastuzumab 6 mg/kg IV. The first doses of trastuzumab and tesevatinib are administered in the clinic on Study Day 1. Subsequent doses of tesevatinib are to be taken on an outpatient basis for the remainder of each 21-day cycle. During Cycle 1, subjects are to be returned to the clinic for weekly safety and tolerability assessments.

Tumor response, both in the central nervous system (CNS) and peripheral to the CNS, is to be assessed after the second cycle of treatment and then at the end of every 2 cycles of treatment thereafter. Subjects are to be treated until disease progression or the subject experienced unacceptable toxicity. Subjects who demonstrated tumor progression are to stop study drug and followed for survival. All subjects discontinuing tesevatinib therapy are to be followed for survival.

Safety assessments include adverse event monitoring, electrocardiograms (ECGs), laboratory testing, physical examinations, vital signs, and pregnancy testing.

An End-of-Treatment visit is to be conducted as soon as possible after the subject's last dose of study drug. This could occur at the visit when disease progression is diagnosed. Subjects are to be followed for disease progression and survival.

A follow-up visit planned for 30 days (± 5 days) after the last dose of study drug assessments is to include collection of AE (Adverse Event) and concomitant medication data. This visit could occur prior to 30 days if a new therapy is started within 30 days of last dose of study drug.

For long-term follow-up, subjects are to be contacted by telephone every 8 weeks to assess survival status and any subsequent anti-cancer treatment.

The duration of treatment for subjects with tesevatinib in combination with trastuzumab is planned until the subject experiences disease progression or unacceptable toxicity.

[Note: Changes to the Planned Analysis: The study, planned to include a Phase 2a expansion in which approximately 50 subjects would have received tesevatinib at the MTD dose determined in Phase 1b, was terminated early. Although some patients had prolonged stable disease in the study, no clear treatment responses were observed. The sponsor decided to suspend the study while gathering additional data from other tesevatinib oncology studies. The study was subsequently terminated early because the sponsor stopped evaluations of tesevatinib as a treatment for HER2-positive metastatic breast cancer.]

ELIGIBILITY:
Inclusion Criteria

Subjects will be included if they meet the following criteria:

1. Female ≥ 18 years old.
2. Females with histologically or cytologically confirmed HER2-positive breast cancer. HER2 positive is defined as 3+ staining by immunohistochemistry, or HER2 gene amplification by fluorescent in situ hybridization (FISH) or silver in situ hybridization (SISH) with HER2/CEP17 ratio ≥ 2.0.
3. Metastatic disease that has progressed on previous therapy or previous therapy was not tolerated.
4. Subjects in the Phase 1b portion of the study and in Group 1 and Group 3 of the Phase 2a portion of the study may have received any number of prior therapies for breast cancer. Subjects in Group 2 of the Phase 2a portion of the study may have received up to 3 lines of therapy in the metastatic setting (not including adjuvant or neoadjuvant therapy).

   1. Previous therapies must have included trastuzumab, pertuzumab, and trastuzumab emtansine. However, subjects starting initial systemic therapy for HER2-positive breast cancer prior to June 2012, when pertuzumab was approved for initial treatment of patients with HER2-positive breast cancer, are not required to have had pertuzumab.
   2. If the subject has ER+ breast cancer, prior therapy must have included at least 1 hormonal therapy.
   3. Subjects with asymptomatic brain metastases found on screening MRI may be entered into Phase 1b or into Group 2 of the Phase 2a without prior radiation therapy to the brain. Subjects with minimally symptomatic brain metastases found on screening MRI may be entered into Phase 1b or into Group 2 of the Phase 2a without prior radiation therapy to the brain if they do not require immediate surgical or radiation therapy in the opinion of the treating investigator and in the opinion of a radiation therapy or neurosurgical consultant.
   4. Subjects with brain metastases that are progressing in the brain after radiation therapy are eligible for enrollment in both Phase 1b and Group 1 of the Phase 2a, provided that there has been no further local therapy for the progressing brain metastases. These subjects must have previously received trastuzumab, pertuzumab (if received initial systemic therapy for HER2-positive breast cancer prior to June 2012 when pertuzumab was approved for initial systemic therapy of HER2-positive, metastatic breast cancer), and trastuzumab emtansine.
   5. Subjects with leptomeningeal metastases may or may not have brain metastases. When brain metastases are present, they do not need to have progressed after radiation therapy.
5. Subjects with disease progression in the brain after prior brain radiation therapy may have extra-CNS metastases in any location or may have no extra-CNS metastases.
6. At least 1 measurable breast cancer lesion that is ≥ 10 mm in one dimension (or

   ≥ 15 mm in shortest axis for lymph nodes) by spiral CT scan or by brain MRI. All brain metastases should be evaluated by T1-weighted, gadolinium-enhanced magnetic resonance imaging (MRI). Subjects with leptomeningeal metastases (Group 3) are not required to have measurable disease but must have cytologic confirmation of leptomeningeal disease.
7. Trastuzumab therapy and hormonal therapy for breast cancer treatment started prior to study entry may be continued. However, previous chemotherapy (including antibodies other than trastuzumab) for breast cancer treatment must have been discontinued at least 14 days before the start of study treatment. Surgical procedures other than port placement must have been performed at least 14 days prior to the start of study treatment. Subjects must have recovered from the reversible effects of prior breast cancer treatments, including surgery and radiation therapy (excluding alopecia).
8. No increase in corticosteroid dose during the week prior to screening brain MRI.
9. No history of another malignancy in the past 5 years, except treated non-melanoma skin cancer or superficial bladder cancer or carcinoma-in-situ of the cervix.
10. ECOG (Eastern Cooperative Oncology Group) status of ≤ 1 (see Appendix C). However, subjects in Group 3 (leptomeningeal metastases) require ECOG status of ≤ 2.
11. Adequate organ and bone marrow functions as follows: (a) Serum creatinine ≤ 1.5 mg/dL; (b) total bilirubin ≤ 1.5 × upper limit of normal (ULN); (c) alanine aminotransferase and aspartate aminotransferase ≤ 3× ULN; (d) white blood cell count > 3000/mm^3; (e) absolute neutrophil count ≥ 1500/mm^3; (f) platelet count > 100,000/mm^3; and (g) hemoglobin > 8 g/dL
12. Serum potassium and magnesium levels within normal limits (WNL).
13. Cardiac ejection fraction WNL as measured by echocardiogram, as long as lower limit of normal (LLN) at the institution is ≥ 50%.
14. No coexisting medical problems of sufficient severity to limit compliance with the study.
15. Willing and able to sign written informed consent and be able to comply with the study protocol for the duration of the study.
16. Women of childbearing potential (ie, menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test). Sexually active women of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes: (a) Intrauterine Device (IUD) plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus 1 barrier method; (c) 2 barrier methods where effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.

Exclusion Criteria

A subject who meets any of the following criteria is ineligible for entry into the study:

1. Any concurrent therapy for breast cancer other than the specified treatment in this study. Concurrent treatment with bisphosphonates or denosumab is allowed, if started prior to the start of tesevatinib administration.
2. Cerebrospinal fluid (CSF) cytology positive for malignant cells or symptomatic leptomeningeal carcinomatosis in the Phase 1b portion of the study. Note: In Group 3 of the Phase 2a portion of the study, subjects are required to have CSF cytology positive for malignant cells.
3. Taking any medication known to inhibit the CYP3A4 isozyme or any drugs that are CYP3A4 inducers (including phenytoin), or any drugs associated with torsades de pointes or known to prolong the QTc(f) interval, including anti-arrhythmic medications within 2 weeks prior to Day 1 of treatment in the study. A stable regimen (≥ 4 weeks) of antidepressants of the SSRI(selective serotonin reuptake inhibitor) class is allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline, and fluoxetine).
4. Has evidence of active heart disease such as myocardial infarction within the 3 months prior to study entry; symptomatic coronary insufficiency or heart block; congestive heart failure; moderate or severe pulmonary dysfunction.
5. History of torsades de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first degree block, being PR(partial response) interval only), or congenital long QT syndrome. Subjects with a history of atrial arrhythmias should be discussed with the medical monitor.
6. Has an active infectious process.
7. Female subject who is pregnant or lactating.
8. Known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body.
9. Has had major surgery without full recovery.
10. Has marked prolongation of QTc interval at screening or baseline (QTc interval > 470 msec) using the Fridericia method of correction for heart rate.
11. History of gastrointestinal (GI) condition that might interfere with drug absorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09-13 (Actual); Study Completion 2015-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - San Juan Oncology, Farmington, New Mexico
  - Laura and Isaac Perlmutter Cancer Center @ NYU Langone, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Open-label, ascending-dose
Groups:
- Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 150 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzumab every 3 weeks
- Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 250 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzumab every 3 weeks
- Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 300 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzumab every 3 weeks
- Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 350 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzumab every 3 weeks
Period: Overall Study
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV
Started | 4 | 3 | 8 | 2
Completed | 0 (Study terminated by sponsor) | 0 (Study terminated by sponsor) | 0 (Study terminated by sponsor) | 0 (Study terminated by sponsor)
Not Completed | 4 | 3 | 8 | 2
Not completed — Death | 1 | 1 | 5 | 1
Not completed — Termination of study by sponsor | 2 | 2 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects entered into study (Safety Population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV | Total
Number analyzed (Participants) | 4 | 3 | 8 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.66) | 50.3 (7.23) | 51.0 (8.80) | 59.5 (2.12) | 49.4 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 8 | 2 | 17
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 8 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 4 | 3 | 7 | 1 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Childbearing potential [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 3 | 0 | 7
  No | 1 | 2 | 5 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Percentage of Subjects With Treatment Emergent Adverse Events (TEAEs) by Severity and/or Relationship to Tesevatinib
Description: Percentage of subjects with at least 1 treatment-emergent adverse event of Grade 3 or greater or relationship with tesevatinib. TEAE grading was by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) where Grade 3 is severe and Grade 4 is life-threatening. TEAEs were considered related to study drug if the investigator assessed them as possibly related, probably related, or related.
Time Frame: Up to 8 months: 1 month (28 days) Screening + 6 months treatment + 1 month follow-up
Population: All subjects who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 300 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg then 6 mg/kg trastuzumab every 3 weeks
- All Patients: Combination of subjects in Cohorts 1, 2, 3, and 4
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV | All Patients
Number analyzed (Participants) | 4 | 3 | 8 | 2 | 17
Participants
  Grade ≥ 3 | 1 | 1 | 5 | 2 | 9
  Related to Tesevatinib | 4 | 3 | 7 | 2 | 16
  Grade ≥ 3 Related to Tesevatinib | 1 | 1 | 2 | 2 | 6

2. Primary Outcome: Safety and Tolerability: Percentage of Subjects With Serious Adverse Event (SAE) Related to Tesevatinib
Description: Percentage of subjects with at least 1 serious adverse event considered related to study drug. SAEs were considered related to tesevatinib drug if the investigator assessed them as possibly related, probably related, or related.
Time Frame: Up to 8 months: 1 month (28 days) Screening + 6 months treatment + 1 month follow-up
Population: All subjects who received at last 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV | All Patients
Number analyzed (Participants) | 4 | 3 | 8 | 2 | 17
Participants | 0 | 1 | 2 | 1 | 4

3. Secondary Outcome: Pharmacokinetics (PK): Mean Serum Cmax After 1 Cycle of Treatment With Tesevatinib + Trastuzumab
Description: The mean of the maximum serum concentration (Cmax) for the combination of tesevatinib and trastuzumab after 1 cycle (Cycle 2 Day 1).
Time Frame: PK samples taken pre-dose, and 1, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: Subjects who completed at least 1 cycle of study drug and had PK (pharmacokinetics) measurements performed on Cycle 2 Day 1. Stratified by tesevatinib dose level, not by initial 8 mg/kg trastuzumab dosing level, i.e., 150 mg tesevatinib PO (by mouth) QD(once daily) / 6 mg/kg trastuzumab IV every 3 weeks. Note: Subjects in Cohort 350 mg tesevatinib received only 8 mg/kg trastuzumab and so were not included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 7
ng/mL | 276 (84.4) | 614 (261) | 394 (177)

4. Secondary Outcome: Pharmacokinetics: Median Serum Tmax After 1 Cycle of Treatment With Tesevatinib + Trastuzumab
Description: The median time of the maximum serum concentration (Tmax) for the combination of tesevatinib and trastuzumab after 1 cycle (Cycle 2 Day 1)
Time Frame: PK samples taken pre-dose, and 1, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: Subjects who completed at least 1 cycle of study drug and had PK measurements performed on Cycle 2 Day 1. Stratified by tesevatinib dose level, not by initial 8 mg/kg trastuzumab dosing level, i.e., 150, 250, and 300 mg tesevatinib with 6 mg/kg trastuzumab. Note: Subjects in Cohort 350 mg tesevatinib received only 8 mg/kg trastuzumab and so were not included in this analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 7
hours | 4.00 [3.97 to 4.00] | 5.98 [4.05 to 8.00] | 6.00 [3.93 to 8.00]

5. Secondary Outcome: Pharmacokinetics: Mean Serum AUC(0-t) (Area Under Curve) of Treatment With Tesevatinib + Trastuzumab
Description: The mean area under the concentration-time curve during the period from 0 to a given time point 't' in the tesevatinib 150 mg QD, 250 mg QD, and 300 mg QD cohorts.
Time Frame: PK samples taken pre-dose, and 1, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: Subjects who completed at least 1 cycle of study drug and had PK measurements performed on Cycle 2 Day 1. Stratified by tesevatinib dose level, not by initial 8 mg/kg trastuzumab dosing level, i.e., 150, 250, and 300 mg tesevatinib with 6 mg/kg trastuzumab. Note: Subjects in Cohort 350 mg tesevatinib received 8 mg/kg trastuzumab and so were not included in this analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 7
hr*ng/mL | 5120 (1530) | 13000 (5750) | 8200 (3390)

6. Secondary Outcome: Pharmacokinetics: Mean AR Cmax After 1 Cycle of Treatment With Tesevatinib + Trastuzumab
Description: The mean of the arithmetic mean accumulation ratio (AR) of the maximum concentration of tesevatinib. The AR is defined as:
  Cmax for Cycle 2 divided by Cmax of Cycle 1.
Time Frame: PK samples taken pre-dose, and 1, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: Subjects who completed at least 1 cycle of study drug and had PK measurements performed on Cycle 2 Day 1. Stratified by tesevatinib dose level, not by initial 8 mg/kg trastuzumab dosing level, i.e., 150, 250, and 300 mg tesevatinib with 6 mg/kg trastuzumab. Note: Subjects in Cohort 350 mg tesevatinib only received 8 mg/kg trastuzumab and so were not included in this analysis.
Measure: Mean (Standard Deviation); unit: ratio (no units)
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 7
ratio (no units) | 3.46 (1.11) | 3.38 (0.993) | 2.21 (1.38)

7. Secondary Outcome: Pharmacokinetics: Mean AR AUC(0-24hr) After 1 Cycle of Treatment With Tesevatinib + Trastuzumab
Description: The mean of the arithmetic mean accumulation ratio (AR) of the area under the concentration-time curve from 0 to 24 hours. The AR is defined as:
  AUC(0-24hr) for Cycle 2 divided by AUC(0-24hr) for Cycle 1.
Time Frame: PK samples taken pre-dose, and 1, 2, 4, 6, 8, and 24 hours post-dose on Cycle 1 Day 1 and Cycle 2 Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio (no units)
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV
Number analyzed (Participants) | 3 | 3 | 7
ratio (no units) | 4.04 (0.762) | 4.23 (1.17) | 2.80 (1.33)

ADVERSE EVENTS:
Time Frame: Assessed up to 8 months: 1 month screening + 6 months treatment + 1 month follow-up
Description: The Medical Dictionary of Regulatory Activities Summary of Classifications and Preferred Terms was used to describe AEs.
  The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE; Version 4.03) was used for grading toxicities. Serious adverse events included those with Grade 4, life-threatening.
Groups:
- Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 150 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzunab every 3 weeks
- Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV: Tesevatinib 250 mg orally administered once daily in combination with Trastuzumab IV 8 mg/kg initially then 6 mg/kg trastuzunab every 3 weeks
Arm/Group | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV | All Patients
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/3 | 5/8 | 1/2 | 8/17
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 5/8 | 1/2 | 7/17
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 8/8 | 2/2 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV (N=4) | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV (N=3) | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV (N=8) | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV (N=2) | All Patients (N=17)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Brain edema (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Metastases to Central Nervous System (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Blood bilirubin incrased (Investigations) | 0 | 0 | 1 | 0 | 1
Transaminase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Tesevatinib 150 mg PO QD + Trastuzumab 8 mg/kg IV (N=4) | Arm 2: Tesevatinib 250 mg PO QD + Trastuzumab 8 mg/kg IV (N=3) | Arm 3: Tesevatinib 300 mg PO QD + Trastuzumab 8 mg/kg IV (N=8) | Arm 4: Tesevatinib 350 mg PO QD + Trastuzumab 8 mg/kg IV (N=2) | All Patients (N=17)
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 7 | 2 | 14
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 7
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 5
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 1 | 9
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 3 | 1 | 5
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1 | 2
Catheter site erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0 | 1
Face edema (General disorders) | 1 | 0 | 0 | 0 | 1
Influenza-like illness (General disorders) | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 1 | 1 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 2
Blood bilirubin incrased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2 | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Brain edema (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Metastases to Central Nervous System (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Visual field defect (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Anemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.